CLINICAL TRIAL: NCT06455085
Title: RESTORE: REducing Future fractureS and Improving ouTcOmes of fRagility fracturE
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300012444; OFP-2022C3-30386 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis; Osteoporotic Fractures; Fragility Fracture
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care Arm (Active Comparator): Participants will be mailed education materials and encouraged to follow up with their primary care physician.
  Interventions: Behavioral: Enhanced Usual Care Arm
- Augmented-Fracture Liaison Service Arm (Experimental): Participants will be mailed education materials. Participants will also be contacted by patient navigators who will guide participants through the process of getting a Bone Health Clinician appointment.
  Interventions: Behavioral: Augmented-Fracture Liaison Service Arm

INTERVENTIONS:
Behavioral: Augmented-Fracture Liaison Service Arm — Patients are contacted by a patient navigator (serving as the liaison) and referred to a bone health clinician.
  Arms: Augmented-Fracture Liaison Service Arm
Behavioral: Enhanced Usual Care Arm — Patients will be mailed education materials and encouraged to follow up with their primary care physician.
  Arms: Enhanced Usual Care Arm

SUMMARY:
RESTORE tests whether Augmented-FLS, where patients are contacted by a patient navigator (serving as the liaison) and referred to a bone health provider, is better than Enhanced Usual Care, which includes patient and PCP education and activation. We also aim to determine the influence of age, race, ethnicity, sex, poverty level, geographic region, and timing of entry into the trial after a fracture on the effectiveness of the two strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older (no upper age limit)
* Sustained a primary fragility fracture (hip/femur, pelvis, clinical spine, humerus, wrist) in the last 12 months
* Participant must self-identify a regular primary care provider (PCP)
* Participant must provide a mailing address
* Participant must plan to remain geographically proximate (able to travel if necessary) to the site from which they are recruited over the next several months

Exclusion Criteria:

* Exposure to the following medications in the prior 12 months;
* Actonel or Atelvia (risedronate)
* Fosamax or Binosto (alendronate)
* Reclast, Zometa, or Aclasta (zoledronic acid, zoledronate)
* Boniva or Bondronat (ibandronate)
* Aredia (pamidronate)
* Prolia (denosumab)
* Evenity (romozosumab)
* Tymlos (abaloparatide)
* Forteo (teriparatide)
* Natpara (parathyroid hormone)
* Evista (raloxifene)
* Duavee (bazedoxifene-conjugated estrogen)
* Miacalcin (calcitonin)
* Diagnosis of the following medical conditions;
* CKD stage 4 or 5 or on dialysis
* Multiple myeloma
* Addison's disease
* Adrenal insufficiency
* Enrolled hospice care
* Solid organ transplant, or expecting a solid organ transplant
* Bone marrow transplant
* History of metabolic bone disease (except osteoporosis) such as Paget's disease, osteomalacia, osteogenesis imperfecta, or Cushing's disease
* Fractures resulting from severe trauma (e.g. motor vehicle accidents, a fall from 2 feet or higher elevation)
* Pathologic fractures secondary to malignancy or infection
* Scheduled appointment with a bone health specialist
* Participant unable to consent on their own (cognitive impairment, dementia, etc.)
* Currently enrolled in another research study that requires taking medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2634 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of subsequent fracture | 24 months post randomization
  Incidence of fracture 24 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Saag, MD, MSc, Principal Investigator — University of Alabama at Birmingham; Maria Danila, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Florida- Gainesville, Gainesville, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Chicago (UIC), UI Health, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Allina Health Orthopedics/NorthStar Trauma Network, Coon Rapids, Minnesota
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, and ICF will be made available upon request at conclusion of the study and after study scientific reports (e.g. abstracts, journal articles) are published.